CLINICAL TRIAL: NCT00280306
Title: White Matter Fiber Tracking and Assessment of White Matter Integrity in the Cervical Spinal Cord - Pilot Study
Brief Title: White Matter Fiber Tracking and Assessment of White Matter Integrity in the Cervical Spinal Cord
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cervical Spine Research Society (Other)
Responsible Party: Principal Investigator, Henning U. Voss, Associate Professor of Physics in Radiology, Weill Medical College of Cornell University
Other Study IDs: 1-Voss
Record Dates: First submitted 2006-01-17; First posted 2006-01-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Cord Compression
MeSH Terms: conditions — Spinal Cord Compression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: No interventions — No intervention

SUMMARY:
White matter fiber tracking may provide a novel tool to assess the integrity of injured motor tracts in the cervical spine. It provides information about fiber directions which is not given by conventional MRI. White matter fiber tracking in the brain is used at several institutions, including our own medical college, for presurgical planning of tumor excision. We believe that the technical and clinical experience gained for the brain can be applied to fiber tracking in the cervical spine as well.

DETAILED DESCRIPTION:
White matter fiber tracking may provide a novel tool to assess the integrity of injured motor tracts in the cervical spine. It provides information about fiber directions which is not given by conventional MRI. White matter fiber tracking in the brain is used at several institutions, including our own medical college, for presurgical planning of tumor excision. We believe that the technical and clinical experience gained for the brain can be applied to fiber tracking in the cervical spine as well. White matter fiber tracking in the cervical spine has some important clinical applications:

* A better understanding of the relationship between abnormal cervical spinal anatomy and the impact on fiber tracts would be helpful in determining the best treatment for a particular patient. It may be able to define the indication and role of surgical decompression and stabilization based on quantifiable and reproducible data obtained with this new imaging technology.
* It could help the surgeon to determine what type of surgical approach to choose (anterior versus posterior surgery, depending on the degree of compression / impingement on nerve fibers).
* Correlation between quantitative diffusion measures and spinal cord injury may be used in monitoring the response to treatment and may therefore be an important parameter for clinicians to follow.
* White matter fiber tracking may also help to determine the pathophysiology underlying cervical spondylotic myelopathy. Currently, there is a debate as to whether cervical spondylitic myelopathy is caused mainly by compressive narrowing of the spinal canal, which may lead to focal ischemia and tissue injury, or whether excessive motion due to cervical spondylosis results in increased strain and shear of spinal axons resulting in injury (Henderson et al., Neurosurgery 56(5):1101-13, 2005). If the latter is correct one would expect diffusion changes along the course of white matter tracks above and below the spondylotic changes.

We will first study a pool of 15 normal control subjects to refine our data acquisition and postprocessing tools, and to sample quantitative diffusion based data for the normal cervical spine. A second group of subjects will include 10 patients with significant cervical spondylosis and upper extremity radiculopathy without myelopathy. The third group will be 10 patients with cervical spondylosis and signs and symptoms of myelopathy. The two patient groups will allow us to define systematic differences between normal values and values in the injured spine.

The DTI data will be processed using tools for artifact correction first and then tools for rendering T2 weighted images, diffusion weighted images, ADC maps and FA values.

ELIGIBILITY:
Inclusion Criteria:

Normal controls Spinal cord injury

Exclusion Criteria:

N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cervical spinal cord compression
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2005-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Imaging study of white matter in spinal cord; define systematic differences between normal values and values in the injured spine | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henning U Voss, Principal Investigator — Weill Medical College of Cornell
Locations (1):
- Weill Medical College of Cornell, New York, New York, United States